CLINICAL TRIAL: NCT01090167
Title: A Phase I, Open-label, Multi-center Study of Clofarabine (JC0707) in Japanese Patients With Acute Myeloid Leukemia (AML)
Brief Title: A Study of Clofarabine in Japanese Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOAML10508
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clofarabine (Experimental)
  Interventions: Drug: clofarabine

INTERVENTIONS:
Drug: clofarabine — Intravenous, 20 mg/m2, 30 mg/m2, 40 mg/m2
  Other Names: Evoltra, Clolar, JC0707

SUMMARY:
This study is sponsored by Genzyme Japan K.K. The purpose of this study is to assess the safety, tolerability and pharmacokinetics of Clofarabine (JC0707) intravenously administered to Japanese adult patients with newly diagnosed or relapsed/refractory Acute Myeloid Leukemia (AML) at 20, 30, and 40 mg/m2/day on a 5-day dose schedule.

DETAILED DESCRIPTION:
This is a Phase I, open-label, multi-center study of Clofarabine administered to Japanese patients with Acute Myeloid Leukemia (AML) who are relapsed/refractory or elderly untreated AML for whom standard induction chemotherapy is unlikely to be of benefit.

Cohort 1 will receive 20 mg/m2/day of Clofarabine once daily for five consecutive days, Cohort 2 will receive 30 mg/m2/day, and Cohort 3 will receive 40 mg/m2/day. Patients will receive one cycle as a rule. However, if there is evidence of some hematologic response after one cycle of treatment with Clofarabine, patients may receive up to a maximum of three cycles. If patients fail to achieve CR or CRp after two cycles of treatment with Clofarabine, further dosing for such patients should be stopped.

Three patients constituting a cohort will receive Clofarabine and will then be assessed for dose limiting toxicities (DLT) at Cycle 1. If none of these three patients develops DLT, the next cohort will be introduced. If one of them develops DLT, three new patients will be added to the cohort, so that six patients in total are included in the tolerability assessment. In this case, treatment of the next cohort is allowed only in the case the number of patients who develop DLT is still one in this six-patient cohort. If two of the six patients develop DLT, however, the tolerability is ruled out. However, if two DLTs are observed at the 20mg/m2/day dose cohort, new patients will be enrolled at cohort -1 15mg/m2/day; and if no more than one of six patients in the cohort develop DLT, it will be considered as the last cohort for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients having diagnosis of relapsed or refractory Acute Myeloid Leukemia (AML) according to the World Health Organization (WHO) criteria or untreated AML patients (60 years to 74 years) for whom standard induction chemotherapy is unlikely to be of benefit as judged by the investigator (or co-investigator)
* Age at the time of informed consent 20 years up to 74 years; 60 years or older for patients with previously untreated AML
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Be able to comply with the study procedures and follow-up examinations specified in this protocol.
* Hepatic, renal, pancreatic, and cardiac function satisfying the laboratory values criteria

Exclusion Criteria:

* Patients having diagnosis of acute promyelocytic leukemia(APL, French-American-British classification M3 or WHO classification of APL with t(15;17)(q22;q12), (PML/RARA and variants)
* Have had prior hematologic stem cell transplant
* Have had prior external beam radiation therapy to the pelvis
* Have systemic fungal, bacterial, viral, or other infection that cannot be controlled and is exhibiting symptoms related to the infection despite appropriate treatment. In addition, patients must have a temperature less than 38.0 for at least 48 hours prior to the first dose of the study drug.
* Have any other severe concurrent disease that is difficult to control by drug therapies, or have a history of serious organ dysfunction or disease involving the liver, kidney, pancreas, heart, or other organ system that may place the patient at undue risk
* Diagnosis of another malignancy, unless the patient meets none of the following conditions: 1) Any persisting treatment-related adverse events; 2) Less than 180 days of disease-free duration counted during the period from the treatment completion to enrollment; note that the patients meeting any of the following conditions is eligible:
* Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia are eligible for this study if treatment for the condition has been completed.
* Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed.
* Have a prior positive test for HBs antigen or antibody, HBc antibody, HCV antibody, or HIV antigen or antibody; note that the patients who have had treatment of vaccine and positive for HBs antibody is eligible.
* Have a clinically significant arrhythmia at screening or a known family history of QT prolongation. Marked prolongation of QTc interval exceeding 450 msec is considered clinically significant
* Have clinical evidence suggestive of central nervous system (CNS) involvement with leukemia
* Have a Psychiatric disorders that would interfere with consent, study participation, or follow-up
* Have had prior treatment with the study drug
* Have had any other chemotherapy or investigational agent received within 30 days prior to the first dose of the study drug
* If received any chemotherapy or investigational agent prior to this time point, drug-related adverse events must be recovered to the baseline value or Grade 1 or less prior to the first dose of the study drug (except for alopecia, and nail changes).
* Is currently participating in another concurrent investigational protocol
* Are pregnant or lactating.
* Male and female patients who are fertile must agree to use an effective means of birth control to avoid pregnancy during the study period and for six months after the last dose of study drug.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) as determined by Dose Limiting Toxicities (DLTs) | 28 days (1st cycle)
Safety as measured by number of patients with at least one adverse events (incidence) | 50 days
Safety as measured by severity of adverse events | 50 days
Safety as measured by duration of adverse events | 50 days
Safety as measured by causality of adverse events | 50 days
Safety as measured by seriousness of adverse events | 50 days
Safety as measured by type of adverse event | 50 days
Safety as measured by number of deaths | 50 days
Safety as measured by number of serious adverse events | 50 days
Safety as measured by number of patients who discontinue due to adverse events | 50 days
Safety as measured by clinically significant changes in hematology | 50 days
Safety as measured by clinically significant changes in chemistry parameters (i.e. serum chemistry) | 50 days
Pharmacokinetic (PK) parameters (Cmax, Tmax, AUC) | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (6):
- Japan (6):
  - Nagoya Daini Red Cross Hospital, Aichi
  - National Hospital Organization Nagoya Medical Center, Aichi
  - University of Fukui Hospital, Fukui
  - Tokai University Hospital, Kanagawa
  - Jichi Medical University Hospital, Tochigi
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Tokyo